CLINICAL TRIAL: NCT00210912
Title: A Comparison of the Efficacy and Safety of Topiramate Versus Placebo for the Prophylaxis of Chronic Migraine
Brief Title: A Study of the Effectiveness and Safety of Topiramate Versus Placebo for Preventing Chronic Migraine Headaches
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR004684
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Migraine
Keywords: prevention; Migraine; chronic; headache
MeSH Terms: conditions — Migraine Disorders; Bronchiolitis Obliterans Syndrome; Headache | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of topiramate as compared to placebo for the prevention of headaches in patients with chronic migraine. Topiramate has been approved to prevent migraine headaches as well as in the treatment of epilepsy.

DETAILED DESCRIPTION:
Migraine headaches can be disabling and can interfere with work and a person's quality of life. Preventing these headaches before they start is the best option. Topiramate, an anti-seizure medication, has been shown to help prevent migraine headaches from occurring. This is a multicenter, randomized, double-blind, placebo-controlled, parallel group study of patients with chronic migraine. The Pretreatment Phase for the study will last up to 56 days and will consist of 2 study periods: a Screening/Washout Period (Day -56 to Day -29) and a Prospective Baseline Period (28 days). Medications being used to prevent migraines will be stopped for 14 to 28 days prior to the Prospective Baseline Period and for the rest of the study. The Prospective Baseline Period will begin on study Day -28 (Visit 2), and patients will maintain a daily headache record during this period. Those who move forward in the study must have had at least 15 headache days during this period, half of which need to be migraine headache days. Patients who finish the Prospective Baseline Period, who have the required rates of headache, and who continue to meet the remainder of the entry criteria will be randomized (like with the toss of a coin) to 1 of 2 treatment groups: topiramate 100 milligrams per day or placebo. The Double-Blind Phase will last 16 weeks. During the first 4 weeks, patients will titrate up to the topiramate dose of 100 milligrams per day or to the maximum tolerated dose, whichever is less. The next 12 weeks is the maintenance phase where you will continue to take the dose that you were taking at the end of the 4-week titration period. The primary hypothesis of this study is that the mean decrease in the number of migraine/migrainous headache days per month is greater in the topiramate group than in the placebo group and topiramate is generally well-tolerated.

Topiramate 25 milligram tablets, 2 tablets by mouth twice daily, or maximum tolerated dose, whichever is less, for 12 weeks, or 2 placebo tablets twice daily for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic migraine
* >=15 headache days per month in past 30 days
* >= 15 headache days, half of which need to be migraine headaches during the prospective baseline period
* MIDAS test score >= 11 at Visit 1
* In generally good health
* If female, using birth control
* No abnormalities on neurological examination

Exclusion Criteria:

* Failed > 2 adequate trials of migraine prevention medications
* Failed topiramate due to lack of effectiveness or adverse events
* Daily headaches of severe intensity during past 30 days
* Cluster, basilar, ophthalmoplegic, or hemiplegic migraines
* Migraines started after age 50
* Other pain greater than migraine pain
* Use of drugs to treat migraines for > 4 days per week during the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2003-09; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Change in the average number of days per month with migraine or migrainous headache by daily headache record.

SECONDARY OUTCOMES:
Absolute change and % change from baseline in the headache index; change in the average daily and worst daily headache severity; quality of life assessments (MIDAS, MSQ, Physician's/Subject's global assessments of change.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Silberstein SD, Lipton RB, Dodick DW, Freitag FG, Ramadan N, Mathew N, Brandes JL, Bigal M, Saper J, Ascher S, Jordan DM, Greenberg SJ, Hulihan J; Topiramate Chronic Migraine Study Group. Efficacy and safety of topiramate for the treatment of chronic migraine: a randomized, double-blind, placebo-controlled trial. Headache. 2007 Feb;47(2):170-80. doi: 10.1111/j.1526-4610.2006.00684.x. PMID 17300356
- See also: Prophylaxis Chronic Migraine — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=622&filename=CR004684_CSR.pdf